CLINICAL TRIAL: NCT04333602
Title: Screening and Treatment of Asymptomatic Bacteriuria in the First Two Months After Kidney Transplant. Randomized Control Trial
Brief Title: Asymptomatic Bacteriuria in Early Kidney Transplantation Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centenario Hospital Miguel Hidalgo (Other)
Responsible Party: Principal Investigator, Jose Manuel Arreola Guerra, Head of the Research department and Nephrologist, Centenario Hospital Miguel Hidalgo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-R-03
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Asymptomatic Bacteriuria; Kidney Transplant Infection

STUDY DESIGN:
Intervention Model Description: Group 1: Asymptomatic Bacteriuria screening and treatment and Group 2: Asymptomatic Bacteriuria screening and No treatment for AB.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both the patient, the primary doctor and the laboratory worker do not know the result of the culture. Only the doctors in charge of this process know the result and contact the patient directly if they are in the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening and Treatment of Asymptomatic Bacteriruria (Experimental): All patients assigned to this arm will be screen with urine culture: post- bladder catheter removal, three weeks post-transplant and before double-J ureteral stent removal. If we detect asymptomatic bacteriuria specific treatment will be instituted.
  Interventions: Diagnostic Test: Urinary culture and treatment if asymptomatic bacteriuria is detected
- Screening and NO treatment of Asymptomatic Bacteriuria (No Intervention): All patients assigned to this arm will be screen with urine culture: post- bladder catheter removal, three weeks post-transplant and before double-J ureteral stent removal. No treatment will be instituted.

INTERVENTIONS:
Diagnostic Test: Urinary culture and treatment if asymptomatic bacteriuria is detected — Urinary culture: post- bladder catheter removal, three weeks post-transplant and before double-J ureteral stent removal. Based in the assigned group If we detect asymptomatic bacteriuria specific treatment will be instituted or No treatment.
  Other Names: Clinical decision based in the presence of asymptomatic bacteriuria
  Arms: Screening and Treatment of Asymptomatic Bacteriruria

SUMMARY:
Urinary tract infection (UTI) continues to be the leading cause of infection and hospitalization in post-kidney transplant (RT) surveillance. Facts such as immunosuppression, anatomical alterations and catheters are part of the factors that contribute to a high prevalence of this condition. The incidence during the first trimester is highly variable and ranges between 15 and 50 %. This variability often depends on the definition of UTI, which sometimes overlaps with asymptomatic bacteriuria (AB). Currently the indication for treatment of AB is clear in pregnant patients and urological procedures. In post-RT surveillance, the treatment of AB is controversial. The use of Trimetropim Sulfamethoxazole during the first 6 months post RT is currently a recommendation, however new evidence has found the absence of benefit in the treatment of AB. Given the high prevalence of post RT AB and the increase in bacterial resistance, determining the usefulness of searching for and treating post RT AB is a priority in this population. Methodology: Randomized Controlled trial of kidney transplant candidates which will be randomized in the following groups: Group 1 (intervention) where the urine cultures will be analyzed openly, and in the case of asymptomatic bacteriuria, treatment based on the germ and antibiogram will be prescribed. Group 2 will undergo urine cultures at the same post-transplant times, the results will not be known by the clinical team and the participants will not receive treatment in the presence of present AB. Both groups, in the presence of UTI symptoms, will undergo urine culture and receive empirical treatment, which will be adjusted based on an antibiogram. The primary objective is to assess the prevalence of UTI, pyelonephritis, UTI-related hospitalizations, and antimicrobial resistance. As a secondary objective, the germs and associated virulence genes will be analyzed. Surveillance will be carried out for two months after transplantation and the predefined times for the evaluation of the BA will be: after the removal of the urinary catheter, week 3 and after the removal of the ureteral stent (month 2).

DETAILED DESCRIPTION:
I. Background Urinary tract infection (UTI) is the most frequent infectious complication in renal transplant recipients (RTR) during the first year, reaching an incidence from 23% to 75%. (1,2) Asymptomatic bacteriuria (AB) and UTI are associated with graft pyelonephritis, sepsis, acute rejection, and long-term graft dysfunction. (3-5) Recently, recurrent UTI episodes have been reported to be associated with poorer patient and graft survival compared to those without recurrent infection. (6) Risk factors are classified as: patient-related (diabetes mellitus, anatomical abnormalities of the urinary tract) and transplant-related (type of immunosuppression, time of the bladder catheter (UC) and double J stent. (7,8) The recommendations of the clinical guidelines suggest prophylaxis with trimethoprim / sulfamethoxazole (TMP / SMX) 160/800 mg every 24 hr during the first 6 months after kidney transplant (KT) ( 9).

The incidence of UTI in RTR has remained between 30 and 36% despite TMP / SMX antimicrobial prophylaxis (7) in a third-level care center in Mexico City; This high incidence is explained in part by the high resistance rate to TMP / SMX (> 80%) in clinical isolates of Escherichia coli recovered from urine both in Mexico and other regions of the world, a condition that discourages its continued use as a prophylactic agent from UTI. (10-12) Given this problem, a clinical trial of kidney transplant recipients was started, comparing the usual prophylaxis with TMP / SMX vs Phosphomycin 3 grams every 10 days for 6 months. The study was suspended prematurely due to therapeutic futility (19). A new clinical trial was performed using intravenous phosphomycin disodium the day of the transplant, prior to the removal of the bladder catheter and the double J ureteral stent. In this study, the intervention group presented a lower incidence of UTI (7.3 vs. 36.6%, p = 0.001).

In both previously described trials, patients underwent UTI screening by urine culture on specific days. Asymptomatic bacteriuria episodes are treated according to the susceptibility of the germ. This alone represents a strategy to decrease the incidence of UTI. Treatment of AB episodes has clearly not been shown to be beneficial in this group of patients. Recently in a controlled clinical trial no benefit was found in KTR with screening and treatment of AB after the second month of post KT. (14) This study partially supports the recommendations of clinical practice of the American Society of Infectious Diseases, where the systematic scrutiny and treatment of the UTI in kidney transplantation is mentioned as not recommended, however the authors propose possible benefit during the first month after KT. (2) II. Definition of the problem Urinary tract infection is the most frequent infectious complication after KT. The systematic screening and treatment of AB during the first months after transplantation is controversial. Given the increase in bacterial resistance, it is important to limit the exposure of antibiotics in high-risk groups. Various studies have demonstrated the utility of the administration of antimicrobial prophylaxis during the first months after transplantation for the reduction of UTI and AB events. However, these studies and several centers carry out systematic scrutiny of UTI with treatment of episodes of AB. Recently a controlled clinical trial showed that the scrutiny and treatment of AB after the second month after transplantation is not useful.

III. Justification UTI represents the most frequent cause of post kidney transplant infection. AB is highly prevalent during the first months after KT. Its prevalence during the first trimester is high and currently the treatment of AB is not fully justified. Due to the need to avoid the abuse of antibiotics in our setting, it is necessary to evaluate the usefulness of screening and treatment of AB in the first 8 weeks post KT. The Medical Center where the trial will be done, performs an average of 100 to 120 kidney transplants annually, which makes the clinical trial feasible.

IV. Hypothesis The screening and treatment of AB during the first 2 months will reduce the incidence of UTI, pyelonephritis and hospitalizations by 50% (composite outcome).

V. Objectives. To assess the efficacy of AB screening and treatment in KT recipients during the first two months post KT.

To assess the incidence of UTI, pyelonephritis and hospitalizations associated with UTI Assess the prevalence of multi-resistant germs The urine culture samples will be labeled and in case of being positive, the isolated strain will be conserved for the subsequent identification of virulence genes. Said strain will be identified with the record of the study of the patient, in order to know the clinical variables of the time of obtaining said sample.

VIII. Definition of monitoring variables Asymptomatic Bacteriuria: In the case of men, medium stream urine culture with isolation of > 1 x 105 colonies. In the case of women, medium-stream urine culture with isolation of > 1 x 105 colonies (2 cultures), must be the same germ.

Urinary tract infection: Isolation of medium stream urine culture >1 x 104 colonies coupled with symptoms such as fever, dysuria, leukocyturia or positive nitrites. If it is only fever, another infectious focus should be ruled out.

Pyelonephritis: Urinary tract infection coupled with fever, graft pain, systemic inflammatory response, or shock. It should not have another concomitant infection.

X. Sample Size:

Taking into account that UTI events occur on average 30% during the first 3 months after KT if the investigators want to reduce events to 10%. Taking the proportions formula. The sample required to be included is 62 patients per maneuver group.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant candidates scheduled for the procedure

Exclusion Criteria:

* Patients with urological complications that did not have a bladder catheter and/or double J ureteral stent removed during the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic urinary tract infection | Two months
  urinary symptoms associated with positive urine culture
Time to the first symptomatic urinary tract infection | Two moths
  urinary symptoms associated with positive urine culture
Incidence of pyelonephritis or hospitalization related to urinary tract infection | Two months

SECONDARY OUTCOMES:
Bacterial virulence genes related to urinary tract infection | Two moths
  E. Coli and Klebsiella. sp virulence genes will be analysed

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Manuel Arreola, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JR, Bang H, Dadhania D, Hartono C, Aull MJ, Satlin M, August P, Suthanthiran M, Muthukumar T. Independent risk factors for urinary tract infection and for subsequent bacteremia or acute cellular rejection: a single-center report of 1166 kidney allograft recipients. Transplantation. 2013 Oct 27;96(8):732-8. doi: 10.1097/TP.0b013e3182a04997. PMID 23917724
- [Background] Britt NS, Hagopian JC, Brennan DC, Pottebaum AA, Santos CAQ, Gharabagi A, Horwedel TA. Effects of recurrent urinary tract infections on graft and patient outcomes after kidney transplantation. Nephrol Dial Transplant. 2017 Oct 1;32(10):1758-1766. doi: 10.1093/ndt/gfx237. PMID 28967964
- [Background] Sorto R, Irizar SS, Delgadillo G, Alberu J, Correa-Rotter R, Morales-Buenrostro LE. Risk factors for urinary tract infections during the first year after kidney transplantation. Transplant Proc. 2010 Jan-Feb;42(1):280-1. doi: 10.1016/j.transproceed.2009.11.029. PMID 20172330
- [Background] de Souza RM, Olsburgh J. Urinary tract infection in the renal transplant patient. Nat Clin Pract Nephrol. 2008 May;4(5):252-64. doi: 10.1038/ncpneph0781. Epub 2008 Mar 11. PMID 18334970
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597
- [Background] Kawecki D, Kwiatkowski A, Sawicka-Grzelak A, Durlik M, Paczek L, Chmura A, Mlynarczyk G, Rowinski W, Luczak M. Urinary tract infections in the early posttransplant period after kidney transplantation: etiologic agents and their susceptibility. Transplant Proc. 2011 Oct;43(8):2991-3. doi: 10.1016/j.transproceed.2011.09.002. PMID 21996207
- [Background] Origuen J, Fernandez-Ruiz M, Lopez-Medrano F, Ruiz-Merlo T, Gonzalez E, Morales JM, Fiorante S, San-Juan R, Villa J, Orellana MA, Andres A, Aguado JM. Progressive increase of resistance in Enterobacteriaceae urinary isolates from kidney transplant recipients over the past decade: narrowing of the therapeutic options. Transpl Infect Dis. 2016 Aug;18(4):575-84. doi: 10.1111/tid.12547. Epub 2016 Jul 4. PMID 27373698
- [Background] Falagas ME, Kastoris AC, Kapaskelis AM, Karageorgopoulos DE. Fosfomycin for the treatment of multidrug-resistant, including extended-spectrum beta-lactamase producing, Enterobacteriaceae infections: a systematic review. Lancet Infect Dis. 2010 Jan;10(1):43-50. doi: 10.1016/S1473-3099(09)70325-1. PMID 20129148
- [Background] Origuen J, Lopez-Medrano F, Fernandez-Ruiz M, Polanco N, Gutierrez E, Gonzalez E, Merida E, Ruiz-Merlo T, Morales-Cartagena A, Perez-Jacoiste Asin MA, Garcia-Reyne A, San Juan R, Orellana MA, Andres A, Aguado JM. Should Asymptomatic Bacteriuria Be Systematically Treated in Kidney Transplant Recipients? Results From a Randomized Controlled Trial. Am J Transplant. 2016 Oct;16(10):2943-2953. doi: 10.1111/ajt.13829. Epub 2016 May 23. PMID 27088545
- [Background] Nicolle LE, Bradley S, Colgan R, Rice JC, Schaeffer A, Hooton TM; Infectious Diseases Society of America; American Society of Nephrology; American Geriatric Society. Infectious Diseases Society of America guidelines for the diagnosis and treatment of asymptomatic bacteriuria in adults. Clin Infect Dis. 2005 Mar 1;40(5):643-54. doi: 10.1086/427507. Epub 2005 Feb 4. No abstract available. PMID 15714408
- [Background] Magiorakos AP, Srinivasan A, Carey RB, Carmeli Y, Falagas ME, Giske CG, Harbarth S, Hindler JF, Kahlmeter G, Olsson-Liljequist B, Paterson DL, Rice LB, Stelling J, Struelens MJ, Vatopoulos A, Weber JT, Monnet DL. Multidrug-resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. Clin Microbiol Infect. 2012 Mar;18(3):268-81. doi: 10.1111/j.1469-0691.2011.03570.x. Epub 2011 Jul 27. PMID 21793988
- [Background] Bauer MP, Kuijper EJ, van Dissel JT; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases (ESCMID): treatment guidance document for Clostridium difficile infection (CDI). Clin Microbiol Infect. 2009 Dec;15(12):1067-79. doi: 10.1111/j.1469-0691.2009.03099.x. PMID 19929973
- [Background] Arreola-Guerra JM, Rosado-Canto R, Alberu J, Maravilla E, Torres-Gonzalez P, Criollo E, Perez M, Mancilla E, Arvizu M, Morales-Buenrostro LE, Vilatoba-Chapa M, Sifuentes-Osornio J. Fosfomycin trometamol in the prophylaxis of post-kidney transplant urinary tract infection: A controlled, randomized clinical trial. Transpl Infect Dis. 2018 Oct;20(5):e12980. doi: 10.1111/tid.12980. Epub 2018 Sep 10. PMID 30133928
- [Result] Alangaden GJ, Thyagarajan R, Gruber SA, Morawski K, Garnick J, El-Amm JM, West MS, Sillix DH, Chandrasekar PH, Haririan A. Infectious complications after kidney transplantation: current epidemiology and associated risk factors. Clin Transplant. 2006 Jul-Aug;20(4):401-9. doi: 10.1111/j.1399-0012.2006.00519.x. PMID 16842513
- [Result] Parasuraman R, Julian K; AST Infectious Diseases Community of Practice. Urinary tract infections in solid organ transplantation. Am J Transplant. 2013 Mar;13 Suppl 4:327-36. doi: 10.1111/ajt.12124. No abstract available. PMID 23465025
- [Result] Fiorante S, Lopez-Medrano F, Lizasoain M, Lalueza A, Juan RS, Andres A, Otero JR, Morales JM, Aguado JM. Systematic screening and treatment of asymptomatic bacteriuria in renal transplant recipients. Kidney Int. 2010 Oct;78(8):774-81. doi: 10.1038/ki.2010.286. Epub 2010 Aug 18. PMID 20720526
- [Result] Golebiewska JE, Debska-Slizien A, Rutkowski B. Treated asymptomatic bacteriuria during first year after renal transplantation. Transpl Infect Dis. 2014 Aug;16(4):605-15. doi: 10.1111/tid.12255. Epub 2014 Jul 1. PMID 24980847